CLINICAL TRIAL: NCT05666583
Title: The Effect of Art Therapy on Pain, Emesis, Anxiety and Quality of Life in Operated Breast Cancer Patients
Brief Title: The Effect of Art Therapy on Pain, Emesis, Anxiety and Quality of Life, Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Esra Baser Akin, Research Asisstant (Researcher in the clinic), Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-11/15
Record Dates: First submitted 2022-12-09; First posted 2022-12-28 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer,; art therapy; marbling art; music therapy; pain,; emesis,; anxiety; quality of life
MeSH Terms: conditions — Breast Neoplasms; Pain; Vomiting; Anxiety Disorders | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Within the scope of the research, the art of marbling was made by the art expert, accompanied by a total of 5 sessions ney concerts for 10 weeks, with two-week intervals. The art application was made to last 20-30 minutes before the patients received chemotherapy. The scales were administered to the individuals in the intervention groups three times in total.
  Interventions: Other: Art therapy
- Control Group (Experimental): No treatment was applied to the control group. The scales were administered to the individuals in the control groups three times in total.
  Interventions: Other: Art therapy

INTERVENTIONS:
Other: Art therapy — The intervention group is the group in which art therapy is applied. They receive chemotherapy.

SUMMARY:
The research sample consisted of 60 individuals, including the intervention group (n=30) and the control group (n=30), who received treatment at the Oncology Center of Sivas Cumhuriyet University Practice and Research Hospital. Personal Information Form, Pain Intensity Measurement-Visual Analog Scale, Rhodes nausea, vomiting and retching index, Beck Anxiety Inventory, FACT-G Quality of Life Scale were applied to the research data. Toxicity Rating Scale total score was recorded from the patient file. Within the scope of the research, a chemotherapy session for 10 weeks (5 sessions) with an interval of two weeks was made by the art expert of the art of marbling, accompanied by a ney concert. No intervention was made in the control group. Within the scope of the research, scale forms will be applied to both groups in the first interview, in the 3rd and 5th chemotherapy sessions of the patients. The data obtained from the study were uploaded to the SPSS (22.0) program and statistical evaluation was made.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received at least one course of chemotherapy, who have undergone breast surgery, who have not been given art therapy, who have no communication difficulties and no mental problems, who are 18 years of age or older, and who agreed to participate in the study.

Exclusion Criteria:

* Those with cancer stage IV, visual, hearing and communication difficulties, those under the age of 18 and those who wanted to leave the study were not included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale: | It will take 10 weeks to collect data three times after randomization is done. The first measurement of pain will be done in the first week, the second measurement in the fifth week and the third measurement in the tenth week.
  It is a scale used to evaluate the pain experienced by patients. Scale; It contains the numbers "start 0 (no pain)" and "10 (severe pain)" at the other end. The patient marks the level of pain he experiences based on these two values.
The Rhodes index of nausea, vomiting and retching (RINVR) | It will take 10 weeks to collect data three times after randomization is done. The first measurement of nausea, vomiting will be done in the first week, the second measurement in the fifth week and the third measurement in the tenth week.
  They found that the alpha internal consistency coefficient of the Nausea, Vomiting and Regurgitation Index, developed by Rhodes and McDaniel and validity and reliability by Rhodes and McDaniel, ranged from 0.98, and the alpha internal consistency coefficients of the subgroups ranged between 0.83 and 0.99. Each response is scored as 0 = least distress, 4 = most distress. The patient's experience of nausea and vomiting in each of the 8 items is summed up. The highest possible value is 32 and represents the most severe symptom occurrence score.It was adapted to Turkish society by Tan and Genç (2010).
Beck Anxiety Scale (BAI) | It will take 10 weeks to collect data three times after randomization is done. The first measurement of anxiety will be done in the first week, the second measurement in the fifth week and the third measurement in the tenth week.
  Beck et al. (1988) in order to determine the frequency of anxiety symptoms experienced by the individual. The scale is a Likert-type self-assessment scale consisting of 21 items and scored between 0-3. The high total score indicates the high level of anxiety experienced by the person. The score range ranges from 0 to 63. Evaluation of the scale is 0-7 points for no anxiety symptoms, 8-15 for mild anxiety, 16-25 for moderate anxiety, and 26-63 for severe anxiety symptoms.
FACT-G Quality of Life Scale | It will take 10 weeks to collect data three times after randomization is done. The first measurement of quality of life will be done in the first week, the second measurement in the fifth week and the third measurement in the tenth week.
  FACT-G is a quality of life scale. In the Turkish naming of this scale, the abbreviation of the original scale [Functional Assessment of Cancer Therapy- General] (FACT-G) is used. It was developed by Cella et al. in 1993. The Turkish validity and reliability of the scale were performed by Çetiner et al. in 2004. This scale has 4 subgroups consisting of 28 items: physical condition, social life and family status, activity status and emotional state. Total scale score is obtained by summing the scores of all items and subgroup scores are obtained by summing the scores of the items in the subgroup. High scores on the total scale and subgroups suggest that patients' quality of life is also high.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra BAŞER AKIN, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mollaog Lu MC, Mollaog Lu S, Akin EB, Mollaog Lu M, Yanmis S. The Effect of Art Therapy on Pain, Emesis, Anxiety, and Quality of Life in Operated Breast Cancer Patients: Randomized Control Trials. J Integr Complement Med. 2024 Apr;30(4):371-382. doi: 10.1089/jicm.2023.0062. Epub 2023 Oct 12. PMID 37824754